CLINICAL TRIAL: NCT07325929
Title: Online Radical Acceptance Intervention for Social Anxiety Disorder: a Randomized Controlled Trial
Brief Title: Online Radical Acceptance Intervention for Social Anxiety Disorder
Acronym: RA-SAD-001
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 457-25
Record Dates: First submitted 2025-12-02; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Social Anxiety Disorder (SAD)
Keywords: social anxiety disorder; acceptance; emotion regulation; guided self-help; digital intervention
MeSH Terms: conditions — Phobia, Social; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: This is a two-arm parallel randomized controlled trial in which participants are assigned to either a self-guided online Radical Acceptance intervention or an active relaxation skills training control condition. All participants complete the same assessment schedule, and each individual receives only the intervention assigned at random.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical Acceptance (Experimental): Participants will receive an online radical acceptance training based on DBT principles. The intervention consists of six guided exercises delivered over a two-week period, designed to enhance acceptance of distressing internal experiences.
  Interventions: Behavioral: Radical Acceptance
- Relaxation Skills (Active Comparator): Participants will receive an online training in DBT TIPP relaxation skills (Temperature, Intense Exercise, Paced Breathing/Progressive Muscle Relaxation). The intervention includes six guided exercises over two weeks, aiming to rapidly decrease physiological arousal and support emotion regulation under stress.
  Interventions: Behavioral: Relaxation Skills

INTERVENTIONS:
Behavioral: Radical Acceptance — Online DBT-based program focusing on implementing radical acceptance in daily life and coping with socially anxious situations.
  Arms: Radical Acceptance
Behavioral: Relaxation Skills — Online DBT-based program teaching relaxation techniques to achieve rapid physiological down-regulation and improve emotional control.
  Arms: Relaxation Skills

SUMMARY:
The goal of this clinical trial is to learn if a self-guided online Radical Acceptance program helps reduce symptoms of Social Anxiety Disorder. The study will also compare this program to an online relaxation skills program.

The main questions are:

* Does the Radical Acceptance program lower symptoms of Social Anxiety Disorder?
* Is the Radical Acceptance program more helpful than relaxation skills?

Adults with Social Anxiety Disorder will be randomly assigned to one of two online programs. They will complete a baseline learning session and six short home practice sessions over two weeks. Participants will answer surveys about their symptoms and complete brief computer tasks. Researchers will measure changes in social anxiety at several points during the study and again a few weeks and a few months later.

DETAILED DESCRIPTION:
This randomized controlled trial will evaluate a self-guided online Radical Acceptance intervention for adults with Social Anxiety Disorder. The intervention is adapted from Dialectical Behavior Therapy (DBT) and is designed to help individuals notice and accept difficult thoughts and feelings that arise during social situations. The study will compare this program with an active control condition that provides training in relaxation skills, also adapted from DBT, which focus on physiological strategies for reducing acute emotional arousal.

The study will enroll 100 adults diagnosed with Social Anxiety Disorder. All study activities take place online. After eligibility is confirmed through structured diagnostic interviews, participants will complete a baseline learning session followed by six home practice sessions delivered over a two-week period. Participants in both conditions will receive culturally adapted video-based training followed by a brief debriefing to ensure understanding and correct application of the assigned skill.

The trial is designed to examine changes in social anxiety symptoms over time and to compare the effects of Radical Acceptance and relaxation skills training. In addition to symptom outcomes, the study will assess several proposed mechanisms of change. These mechanisms include interpretation bias and emotion regulation flexibility measured through behavioral tasks, as well as experiential avoidance, rumination, and difficulties in emotion regulation measured through self-report instruments. Mechanism assessments will be completed at baseline and after the fourth practice session. Participants will also report their momentary positive and negative emotions before and after each practice session.

Recruitment will occur through online advertisements. Screening includes an online questionnaire followed by a telephone interview and a video-based diagnostic assessment using the ADIS-5 and selected DIAMOND modules, administered by trained graduate students. Eligible individuals will provide informed consent for both the assessment session and the intervention phase of the study.

Participants will be randomly assigned by an automated algorithm to one of the two study conditions. All assessments and intervention procedures will be completed remotely. The study includes follow-up assessments at three weeks and three months after the intervention to evaluate the stability of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* Score > 9 on Mini-SPIN
* Positive responses in brief phone screening
* Eligibility confirmed in Zoom interview using ADIS
* Native Hebrew speakers
* Having regular access to a computer.

Exclusion Criteria:

* Changes in psychiatric medication in the past 3 months
* Current or past diagnosis of bipolar disorder
* Current or past diagnosis of schizophrenia
* Current or past diagnosis of PTSD
* Current or past diagnosis of substance use disorder
* History of traumatic brain injury (TBI)
* Previous experience with Dialectical Behavior Therapy (DBT)
* Currently receiving psychotherapy specifically targeting social anxiety

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Liebowitz Social Anxiety Scale | baseline, after session 4 (~1 week), 2 weeks (end of treatment), 3-week follow-up, 3-month follow-up
  Change in social anxiety symptoms using the self-report Liebowitz Social Anxiety Scale (LSAS). In this questionnaire, participants are asked to respond to 24 social situations by marking how much they feel fear in each situation (anxiety subscale) and to which extent they will avoid this situation (avoidance subscale) on a 0-3 Likert scale. This measure ranges 0-144; higher scores indicate greater social anxiety severity.

SECONDARY OUTCOMES:
Generalized Anxiety Disorder-7 | baseline, after session 4 (~1 week), 2 weeks (end of treatment), 3-week follow-up, 3-month follow-up
  Change in social anxiety symptoms using the self-report Generalized Anxiety Disorder-7 (GAD-7). Participants rate how frequently they have been bothered by each symptom over the past two weeks using a 4-point Likert scale (0-3). This questionnaire ranges 0-21; higher scores indicate greater anxiety severity.
Patient Health Questionnaire-9 | Time Frame: baseline, after session 4 (~1 week), 2 weeks (end of treatment), 3-week follow-up, 3-month follow-up
  Change in depressive symptoms will be assessed using the Patient Health Questionnaire-9 (PHQ-9). Respondents report how often they have experienced each symptom over the past two weeks using a 4-point Likert scale (0-3). This questionnaire ranges 0-27; higher scores indicate greater depressive symptom severity.

OTHER OUTCOMES:
Word-sentence association task | baseline, after session 4 (~1 week)
  Change in interpretation bias will be evaluated using a word-sentence association task (WSAP). The dependent variable is the proportion of trials in which participants selected the negative interpretation, with higher proportions indicating a stronger negative interpretation bias.
Emotional faces task | baseline, after session 4 (~1 week)
  Change in interpretation bias using a computerized task with facial emotion stimuli. In this task, two dependent measures were derived: the proportion of trials in which participants accurately identified the intended emotional expression for each emotion category (e.g., correctly labeling a happy face as positive).
Emotion regulation flexibility task | baseline, after session 4 (~1 week)
  Change in emotion regulation flexibility as measured by a computerized experimental task. The dependent variables will include the number of trials in which participants chose to use cognitive reappraisal, and the average level of negative affect reported following trials in which reappraisal was selected, serving as an index of implementation success.
Brief Experiential Avoidance Questionnaire | baseline, after session 4 (~1 week)
  Change in experiential avoidance as measured by the Brief Experiential Avoidance Questionnaire (BEAQ). Items are rated on a 6-point Likert scale (1-6). scores range 15-90; with higher scores indicate greater experiential avoidance.
Ruminative Responses Scale | baseline, after session 4 (~1 week)
  Change in rumination as measured by the Ruminative Responses Scale (RRS).Participants rate each statement on a 4-point Likert scale ranging from 1 ("almost never") to 4 ("almost always"), indicating how frequently they respond to feelings of sadness or low mood in the described manner. The RRS yields a total rumination score as well as three subscales representing distinct aspects of ruminative thought: (1) Brooding, (2) Reflection, and (3) Depressive rumination. Higher scores indicate greater rumination.
Positive and Negative Affect Schedule | Before and after each of the six practice sessions: ~day 2, 4, 6, 8, 10, 12
  Change in positive and negative emotions by selected items from the Positive and Negative Affect Schedule (PANAS). We selected the 12 most relevant items from the pool for our study, assessing basic negative and positive emotion scales such as fear, sadness, hostility, joviality, self-assurance and attentiveness. Each item will be scored on a 4-point Likert-scale ranging from 1-5. Higher ratings indicate stronger emotional reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Noam Weinbach, PhD, Principal Investigator — School of Psychological Sciences, University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will depend on ethical approvals, institutional policies, and participant privacy considerations. A final decision about IPD sharing will be made after study completion.